CLINICAL TRIAL: NCT02091479
Title: Randomized Assay Evaluating the Risk/Benefit of Early Versus Late Resumption of Anticoagulation in Patients With Major, Non-trauma Related Hemorrhage Occurring While on Anticoagulant Treatment for a High Risk of Thrombosis.
Brief Title: Early Versus Late Resumption of Anticoagulation in Patients With Both High Thrombosis Risk and Major HEmoRrhage
Acronym: RATHER
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: inclusion rate insufficient
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1108097; 2012-000286-21 (EudraCT Number)
Record Dates: First submitted 2014-03-07; First posted 2014-03-19 (Estimated); Last update posted 2016-03-10 (Estimated); Status verified 2016-03

CONDITIONS: Major hæmorrhage
Keywords: hæmorrhage, thrombosis
MeSH Terms: conditions — Thrombosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- UFH Early group (Experimental): anticoagulant (UFH or LMWH) reintroduction at 48h to 72h after hemorrhage
  Interventions: Drug: UFH Early group
- UFH Late group (Active Comparator): anticoagulant (UFH or LMWH) réintroduction 120h to 144h after hemorrhage
  Interventions: Drug: UFH Late group

INTERVENTIONS:
Drug: UFH Early group — Either curative dose, intravenous unfractionated heparin (UFH) so as to reach an anti-Xa activity between 0.3 and 0.7 IU/mL, lengthening the activated prothrombin time as determined by each centre according to the treatment area (depending on the coagulometer and reactants).
  Or low-molecular-weight, curative dose, subcutaneous heparin (LMWH) so as to reach an anti-Xa activity corresponding to treatment areas as determined for each type of molecule (about 0.5 to 1 anti-Xa IU for most LMWHs, administered via 2 daily injections, and about 0.5 to 1.5 anti-Xa IU for tinzaparin, 1 injection daily).
  Arms: UFH Early group
Drug: UFH Late group — Either curative dose, intravenous unfractionated heparin (UFH) so as to reach an anti-Xa activity between 0.3 and 0.7 IU/mL, lengthening the activated prothrombin time as determined by each centre according to the treatment area (depending on the coagulometer and reactants).
  Or low-molecular-weight, curative dose, subcutaneous heparin (LMWH) so as to reach an anti-Xa activity corresponding to treatment areas as determined for each type of molecule (about 0.5 to 1 anti-Xa IU for most LMWHs, administered via 2 daily injections, and about 0.5 to 1.5 anti-Xa IU for tinzaparin, 1 injection daily).
  Arms: UFH Late group

SUMMARY:
In patients with a high thromboembolic risk, withdrawing anticoagulant treatment is recommended in some situations, including when major hæmorrhage occurs. But withdrawing treatment can be risky. In patients on a curative dose of anticoagulant medicine, treatment withdrawal heightens the risk of thromboembolic events occurring, with potentially major consequences. For instance, mechanical valve thrombosis is fatal in 15% of patients. Resumption of anticoagulation is therefore critical in patients at high risk for thromboembolic events.

However, in these patients having presented major hæmorrhage, resumption of anticoagulation heightens the risk of hæmorrhage recurrence. This risk is even higher when the original hæmorrhage was not accessible via surgical, endoscopic or endoluminal hemostasis.

As far as investigators know, there is no data in the literature to rely on when the major hæmorrhage is not accessible via hemostatic intervention and the risk of thrombosis is high. When confronted with patients who need anticoagulation but have a high risk of hæmorrhage recurrence, the question of when treatment should be resumed has not been resolved. This is why investigators propose to conduct a randomised comparative study to evaluate two treatment strategies - early resumption (H48 to H72) versus late resumption (H120 to H144) of anticoagulation.

MAIN OBJECTIVE: The main objective of the present study is to evaluate in terms of bleeding risk, thrombosis risk and mortality at one month, the effect of early vs. late resumption of anticoagulation in patients having presented with serious hæmorrhage while on curative-dose anticoagulants and facing a high thromboembolic risk.

DETAILED DESCRIPTION:
STUDY DESIGN: This is a comparative, randomised, open study assessing after 1 month and 3 months the effect of early (H48 to 72) versus late (H120 to 144) resumption of anticoagulation in patients presenting with serious bleeding while on anticoagulants (excluding intracerebral bleeding) and with a thromboembolic risk evaluated as high (except mitral prostheses). The accumulated frequency of major hæmorrhage, thromboembolic events and deaths should be 26% in case of early resumption and 15% in case of late resumption, i.e. a relative risk reduction of 43%. Based on this hypothesis, to obtain 80% power with two-sided α being 5%, each group should include 208 patients, for a total of 416 patients.

EVALUATION CRITERIA: The main criteria in this study will be the accumulated one-month incidence of hæmorrhage recurrence, thromboembolic complications and deaths. It is a combined criterion associating:

* Fatal hæmorrhage proven by autopsy or sudden deaths in a clinical context strongly suggestive of hæmorrhage
* Fatal thromboembolic events proven by autopsy or imagery or sudden deaths in a clinical context strongly suggestive of thrombosis
* Any clinically significant hæmorrhage leading to temporary (> 24 hours) or permanent withdrawal of anticoagulant treatment
* Any symptomatic thromboembolic event in any territory, proven by imagery or surgery

These events will be validated by a committee for the validation of critical events blind to the date of anticoagulant treatment resumption. The secondary evaluation criteria will be symptomatic hæmorrhages, fatal or not, symptomatic thromboembolic incidents, fatal or not, and mortality at 1 month and 3 mont

ELIGIBILITY:
Inclusion Criteria:affiliated with or a beneficiary of a social security category

* age > 18 years old
* with major bleeding (ISTH) and highs thrombosis risk (ACCP 2008)
* having signed the inform consent form

Exclusion Criteria:

* intracranial bleeding
* artificial heart valves
* bleeding with hemostatic surgical
* low and moderate thrombosis risk
* INR>1.2
* hemodynamic instability contra-indication to HBPM or HNF treatment
* With previous history of HIT (heparin Inducted thrombopenia)
* patient who need antiaggregant treatment before anticoagulant treatment
* Hæmoglobin count < 8 g/dl or patients with hæmoglobin count < 10 g/dl combined with acute coronary syndrome or proven heart failure
* pregnant
* Polytraumatism
* with curatif heparin before randomisation

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2013-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
The main criterion in this study is the cumulated incidence of mortality, hæmorrhage recurrence and thromboembolic complications at 1 month | The main criterion in this study is the cumulated incidence of mortality, hæmorrhage recurrence and thromboembolic complications at 1 month
  Fatal hæmorrhage proven by autopsy or sudden deaths in a clinical context strongly suggestive of hæmorrhage,
  * Fatal thromboembolic events proven by autopsy or imagery or sudden deaths in a clinical context strongly suggestive of thrombosis,
  * Any clinically significant hæmorrhage leading to temporary (> 24 hours) or permanent withdrawal of anticoagulant treatment,
  * Any symptomatic thromboembolic event in any territory, proven by imagery or surgery,
  * Any heart valve thrombosis or any intracavitary thrombus spotted by transesophageal echocardiogram performed systematically in patients with mechanical prosthesis or valvular rheumatic heart disease or AF.

SECONDARY OUTCOMES:
-We will evaluate the risk/benefit balance of early versus late resumption of anticoagulant treatment, | We will evaluate at 1 month and at 3 monthsthe risk/benefit balance of early versus late resumption of anticoagulant treatment
  * Fatal hæmorrhages proven by autopsy or imagery or sudden deaths in a clinical context strongly suggestive of hæmorrhage,
  * Fatal thromboembolic events proven by autopsy or imagery or sudden deaths in a clinical context strongly suggestive of thrombosis,
  * Any clinically significant hæmorrhage leading to temporary (> 24 hours) or permanent withdrawal of anticoagulant treatment,
  * Any symptomatic thromboembolic event in any territory, proven by imagery or surgery,
  * Any heart valve thrombosis or any intracavitary thrombus spotted by transesophageal echocardiogram performed systematically in patients with mechanical prosthesis or valvular rheumatic heart disease or AF.

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Tardy, MD phD, Principal Investigator — CHU SAINT-ETIENNE
Locations (2):
- France (2):
  - CHU de Saint-Etienne, Saint-Etienne, Saint-etienne
  - Service d'Urgences et de Réanimation Medicale, CHU de Saint-Etienne, Saint-Etienne